CLINICAL TRIAL: NCT02082236
Title: Pharmacokinetics of Sufentanil Sublingual Microtablet 30 mcg and 15 mcg in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SAP101
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: Plasma concentrations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Active Comparator): Sufenta® IV (50 mcg/mL) 30 mcg infused over 1 minute
  Interventions: Drug: Treatment Arm A: Sufenta®
- Treatment B (Experimental): Single dose of SSM 30 mcg
  Interventions: Drug: Treatment B: Sufentanil SSM 30 mcg
- Treatment C (Experimental): 2 consecutive doses of SSM 15 mcg administered 20 minute apart
  Interventions: Drug: Treatment C: SSM 15 mcg
- Treatment D (Experimental): 12 consecutive doses of SSM 30 mcg administered 1 hour apart
  Interventions: Drug: Treatment D: SSM 30 mcg

INTERVENTIONS:
Drug: Treatment Arm A: Sufenta® — Sufenta® intravenous (IV) (50 mcg/mL) 30 mcg infused over 1 minute
  Arms: Treatment A
Drug: Treatment B: Sufentanil SSM 30 mcg — single-dose SSM 30 mcg
  Arms: Treatment B
Drug: Treatment C: SSM 15 mcg — 2 consecutive doses of SSM 15 mcg administered 20 minutes apart
  Arms: Treatment C
Drug: Treatment D: SSM 30 mcg — 12 consecutive doses of SSM 30 mcg administered 1 hour apart
  Arms: Treatment D

SUMMARY:
The purpose of this study is to establish the single and multiple-dose pharmacokinetics (PK) of sublingual administration of the Sufentanil Sublingual Microtablet (SSM) 30 mcg and compare the pharmacokinetics of a single dose of SSM 30 mcg to 2 doses of SSM 15 mcg administered 20 minutes apart.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking male or female subjects
2. Aged between 18 and 45 years inclusive
3. Subjects must have Body Mass Index (BMI) between 18 and 30, inclusively.

Exclusion Criteria:

1. Subjects who are taking over-the-counter medication (except for single dose multi-vitamin supplements or acetaminophen of less than 2 g/day) within 14 days prior to start of sufentanil dosing prescription medications or over the counter (OTC) medications
2. Female subjects who are pregnant
3. Subjects with chronic obstructive pulmonary disease, sleep apnea, or other significant respiratory disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve | 9 days, not including a 30 day screening window
  Area under the plasma concentration time curve

OTHER OUTCOMES:
C max | 9 days
  Maximum plasma concentration
T max | 9 days
  Time to reach maximum plasma concentration
Context Sensitive Half-Time (CST½) | 9 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K. Willsie, D.O., Principal Investigator — PRA
Locations (1):
- PRA, Lenexa, Kansas, United States